CLINICAL TRIAL: NCT06382805
Title: Comparison of the Effects of Kinesio Tape and High-intensity Laser Therapy on Pain, Grip Strength and Functional Level in Patients with Lateral Epicondylitis: a Randomized Controlled Study.
Brief Title: Comparison of the Effects of Kinesio Tape and High-intensity Laser Therapy in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, abuzer akbaş, PhD student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HasanKU_FTR_AA_02
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Tennis Elbow; Physical Therapy; Kinesiotaping; Laser
MeSH Terms: conditions — Tennis Elbow | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: There are three groups in the study. The groups consist of the control group, kinesio tape group and high intensity laser group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): The physiotherapy program will consist of cold-pack, US, transcutaneous electrical stimulation (TENS) and home exercise program.
  Interventions: Other: Physiotherapy program
- kinesiotaping group (Active Comparator): Kinesio tape application will be applied to the kinesio tape group in addition to physiotherapy.
  The physiotherapy program will consist of cold-pack, US, transcutaneous electrical stimulation (TENS) and home exercise program.
  Interventions: Other: Physiotherapy program; Other: Kinesio Tape
- high intensity laser therapy group (Active Comparator): High-intensity laser application will be applied to the high-intensity laser group in addition to physiotherapy. The physiotherapy program will consist of cold-pack, US, transcutaneous electrical stimulation (TENS) and home exercise program.
  Interventions: Other: Physiotherapy program; Other: High Intensity Laser therapy

INTERVENTIONS:
Other: Physiotherapy program — The physiotherapy program will consist of cold-pack, US, transcutaneous electrical stimulation (TENS) and home exercise program. Cold-pack will be applied for 15 minutes. Continuous ultrasound will be applied on lateral epicondylitis with a 5-cm ultrasound head at a dose of 1.5W/cm2 for 5 minutes and a frequency of 1-MHZ. TENS application will be performed with the BTL 4000 combination device. TENS will be applied for 20 minutes, increasing the intensity of the current until the patient feels it. The treatment program will last for a total of two weeks, 5 days a week.
Other: Kinesio Tape — The longitudinal muscle technique will be applied from the origin to the insertion of the forearm extensor muscles by a researcher with a Kinesio tape application certificate. In addition, transverse kinesio tape will be applied on the elbow using the fascia correction technique. The treatment program will last for a total of two weeks, 5 days a week.
  Arms: kinesiotaping group
Other: High Intensity Laser therapy — High intensity laser applications will be performed using the BTL-6000 (BTL Company, UK) device. The first 5 sessions will be applied to the painful area for 75 seconds at a dose of 4W 6 J/cm2 (analgesic effect) by making circular movements from the center to the outside. The remaining 5 sessions will be applied to the painful area with linear movements for 12 minutes and 30 seconds at a dose of 6W 100-150 J/cm2 (biostimulation effect). The treatment program will last for a total of two weeks, 5 days a week.
  Arms: high intensity laser therapy group

SUMMARY:
Lateral epicondylitis is a common upper extremity disease that occurs with tenderness in the lateral epicondyle, the common attachment point of the wrist extensor muscles, and pain during resisted wrist extension. The main purpose of treating lateral epicondylitis is to reduce pain and increase functionality, but there is no accepted standard treatment method. The purpose of this study is to compare the effectiveness of kinesio tape and high intensity laser in the treatment of lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis is a common upper extremity disease that occurs with tenderness in the lateral epicondyle, the common attachment point of the wrist extensor muscles, and pain during resisted wrist extension. It is usually a non-inflammatory tendinopathy of the extensor carpi radialis and extensor digitorum comminis. Calcific tendinitis and/or partial tears in the wrist extensor muscles may accompany this condition. It is most common between the ages of 30-60 and its prevalence has been reported as 1-1.7% Although the underlying cause is mostly unknown, activities that involve excessive use of wrist extensors and supinators are thought to be the most important cause of lateral epicondylitis .The main purpose of treating lateral epicondylitis is to reduce pain and increase functionality, but there is no accepted standard treatment method. Non-surgical treatment approaches such as patient education physiotherapy applications, manual therapy, laser therapy, splinting, taping, exercises, massage and local injection, as well as oral or topical nonsteroidal anti-inflammatory drugs are frequently applied. Kinesio tape, which is frequently used in musculoskeletal system injuries, is flexible, mimics skin and has a water-resistant structure. Kinesio tape creates a pumping system by pulling the skin up in the area where it is applied, thus increasing the skin space, increasing blood and lymph circulation, and creating analgesia and proprioceptive sensory input by reducing the pressure on pain receptors . There are scientific studies showing that kinesio tape application reduces pain and increases functionality and grip strength in patients with lateral apicondylitis. It is stated that high-intensity laser treatment can quickly create photochemical and photothermic effects in deep tissue. For this reason, collagen production in tendons is stimulated and can increase blood flow, vascular permeability and cell metabolism. As a result of all these events, tissue healing begins and painful stimuli disappear. It has been shown that high-intensity laser reduces pain and increases functionality and grip strength in patients with lateral epicondylitis. In the literature review, no randomized controlled studies were found comparing high-intensity laser and kinesio tape applications in patients with lateral epicondylitis

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Those who have pain with palpation applied to the lateral epicondyle
* Patients with pain in resisted extension of the wrist and/or middle finger
* Pain during static stretching applied to the wrist while the elbow is extended
* The complaints must last at least three months
* Not having received treatment in the last three months.

Exclusion Criteria:

* Pregnant and breastfeeding women
* History of fracture or surgery in the elbow area
* Detection of calcific tendinitis on plain radiograph of the elbow
* History of neurological disease
* History of osteoporosis, malignancy, hemophilia
* Rheumatoid arthritis and other inflammatory diseases
* Cognitive problem

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Pain Measurement | Pain will be evaluated before treatment, immediately after treatment and 6 weeks after treatment
  Patients' lateral epicondylitis pain intensity will be evaluated with a visual analog scale (VAS). On the visual analog scale, the left end of a 10 cm straight line represents no pain, and the right end represents excruciating pain. The patient will be asked to mark the pain he feels on the VAS scale during the test, and then this value will be measured and recorded with the help of a ruler.
Hand grip strength | Hand grip strength will be evaluated before treatment, immediately after treatment and 6 weeks after treatment
  A standard hand dynamometer (Jamar® Plus + Digital Hand Dynamometer from Patterson Medical, Sammons Preston, Bolingbrook, USA) will be used to measure grip strength. The Jamar dynamometer has high reliability and validity; therefore the device has been considered the gold standard for assessing grip strength. Grip strength evaluation will be performed with patients in a sitting position from a chair. During the test, patients will be asked to position their elbows in 90° flexion and their forearms and wrists in neutral position. The test will be repeated 3 times with one minute intervals and the average of the obtained values will be recorded.
Patient-Rated Tennis Elbow Evaluation | Patient-Rated Tennis Elbow Evaluation will be evaluated before treatment, immediately after treatment and 6 weeks after treatment
  Functional levels of the patients will be assessed with a Patient-Rated Tennis Elbow Evaluation questionnaire. The questionnaire consists of a total of 15 questions evaluating the functional level of patients with lateral epicondylitis in the last week. 5 questions evaluate pain and the other 10 questions evaluate functional level in various tasks. The score for each question is between 0 (best) and 10 (worst). The best score that can be obtained in the section that evaluates functionality is 0, while the worst score is 100.

SECONDARY OUTCOMES:
Pain Sensitivity Measurement | Pain Sensitivity Measurement will be evaluated before treatment, immediately after treatment and 6 weeks after treatment
  Pain sensitivity will be measured with a pressure pain meter (JTECH Medical, Midvale, UT, USA). Measurements will be made by the same researcher under the same conditions. The researcher will press a 1 cm2 probe perpendicularly to the affected lateral epicondyle and the first point where the patient feels pain will be recorded. Measurements will be repeated 3 times and the average of these values will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: abuzer akbas, Principal Investigator — hasan kalyoncu university faculty of health science
Locations (1):
- Adıyaman training and research hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No